CLINICAL TRIAL: NCT03208335
Title: A Phase II Trial Of Rh-Endostatin In Combination With Radiotherapy In The Treatment Of Hepatocellular Carcinoma
Brief Title: Recombinant Human Endostatin(Rh-endostatin) Combine With Radiotherapy in the Treatment of Hepatocellular Carcinoma(HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Vice Director of Department of Radiotherappy, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLAGH-HCC
Record Dates: First submitted 2017-07-02; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: rh-endostatin; radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Endostatins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rh-endostatin combination (Experimental): Continuous intravenous pumping (CIP) recombinant human endostatin(rh-endostatin) 30mg/d, from 5 days before radiotherapy,for 7days,21 per cycle.Standard radiotherapy for HCC is conducted concurrently.Those patients will receive 3-5 cycles rh-endostatin after the radiotherapy is finished,4-6 cycles in all.
  Interventions: Drug: recombinant human endostatin

INTERVENTIONS:
Drug: recombinant human endostatin — The cycles of rh-endostatin's treatment depends on the effect of reaction and tolerance.
  Other Names: rh-endostatin

SUMMARY:
Hepatocellular carcinoma(HCC) is a high malignancy cancer which progress rapidly , and the rates of morbidity and mortality is very high in China. Radiotherapy as a effective treatment is commonly used in unresectable HCC patients. Preclinical models have shown that anti-angiogenesis medicine,such as rh-endostatin, can normalize the tumor vasculature to make it more efficient for oxygen delivery, which can enhance the radiosensitivity subsequently. This study is to evaluate the safety and efficacy of rh-endostatin combined with radiotherapy in the treatment of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma,or radiographic indicative HCC with AFP>250ug/l
* Inoperable and untransplantable,Child-pugh score A or B
* PS score 0-1
* At least one measurable site(diameter >20mm measured by CT or MRI,>10mm measured by helical CT scan.
* No distant metastases
* Life expectancy longer than 3 months
* Willingness and ability to comply the study and signed informed consent.

Exclusion Criteria:

* Not comply the designed treatment or change to other treatment
* Miss follow-up visits or have incomplete follow-up data
* The efficacy will not be assessed if the Patient withdrawal the treatment due to severe adverse events(SAE),but SAE will be recorded.
* Disease progression
* Patients request to withdraw
* Patients with III hematologic or Ⅳ nonhematologic drug related toxicity ,or SAE

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
progress-free survival(PFS) | 18 months
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause

SECONDARY OUTCOMES:
response rate(RR) | 18months
  CR(complete response)+PR(partial response)
clinical benefit rate(CBR) | 24months
  CR+PR+SD(stable disease)
overall survival(OS) | 36 months
  Overall survival was defined as the time from randomization to death from any cause.
adverse event(AE) | 36 months
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause
Quality of life (QOL) | 36months
  A questionnaire with questions referred to simple assessments of physical abilities

CONTACTS AND LOCATIONS:
Overall Officials: Yu Li, MD, Principal Investigator — China PLA hospital
Locations (1):
- Chinese PLA Gereral Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided